CLINICAL TRIAL: NCT06186271
Title: International Active Surveillance Study: Safety of Estrogen Estetrol (E4) Contraceptive Study (INAS-SEECS)
Acronym: INAS-SEECS
Status: Recruiting | Type: Observational
Sponsor: Center for Epidemiology and Health Research, Germany (Other)
Collaborators: Estetra (Industry); Gedeon Richter Plc. (Industry)
Responsible Party: Sponsor
Other Study IDs: ZEG2022_03
Record Dates: First submitted 2023-12-15; First posted 2023-12-29 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-03

CONDITIONS: Contraception
Keywords: Birth control

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- E4/DRSP: E4/DRSP: estetrol/drospirenone
  new users (starters and restarters with at least two months break)
- EE/DRSP: EE/DRSP: ethinyl estradiol/drospirenone
  new users (starters and restarters with at least two months break)
- EE/LNG and EE/NETA and EE/NGM: EE/LNG: ethinyl estradiol/levonorgestrel
  EE/NETA: ethinyl estradiol/norethisterone/norethindrone acetate
  EE/NGM: ethinyl estradiol/norgestimate
  new users (starters and restarters with at least two months break)

SUMMARY:
The combined oral contraceptive (COC) containing estetrol (E4) and drospirenone (DRSP) (E4/DRSP) is a novel oral contraceptive containing a fixed dose of E4 (14.2 mg) and DRSP (3 mg). The proposed study will address post-market requirements for E4/DRSP under section 505(o) in response to the Food and Drug Administration (FDA) request.

The primary objective of the study is to characterize and compare the risks of E4/DRSP with EE/DRSP and E4/DRSP with a pooled cohort of users of EE/LNG, EE/NETA, and EE/NGM combinations (non-DRSP-containing COCs) in a study population of actual users of these preparations under routine clinical practice. The main clinical outcome of interest is VTE.

DETAILED DESCRIPTION:
Rationale and background: The combined oral contraceptive (COC) containing estetrol (E4) and drospirenone (DRSP) (E4/DRSP) is a novel oral contraceptive containing a fixed dose of E4 (14.2 mg) and DRSP (3 mg). E4 is a natural estrogen only produced during pregnancy by the fetal liver. When combined with the progestin DRSP, ovarian activity is suppressed, and there is less impact on hepatic parameters and hemostasis in comparison to combinations of ethinyl estradiol (EE) and levonorgestrel (LNG) or EE and DRSP. The E4/DRSP combination has now received marketing authorization in multiple locations, including the United States of America (USA). The proposed study will address post-market requirements for E4/DRSP under section 505(o) in response to the Food and Drug Administration (FDA) request.

Two co-primary comparisons will be conducted regarding the risk of venous thromboembolism (VTE) and arterial thromboembolism (ATE): new users of E4/DRSP vs. non-DRSP COCs (comprising LNG, norethisterone/norethindrone acetate [NETA] and norgestimate [NGM] in combination with EE) and E4/DRSP vs. other DRSP-containing products (EE/DRSP) among women of reproductive age using COCs primarily for contraceptive reasons. An adequate number of obese women in the US population will be included for analysis. The study will be adequately powered to rule out a 2.0-fold increase in the risk of VTE for both the E4/DRSP vs. non-DRSP COCs, and the E4/DRSP vs. EE/DRSP COCs analyses.

Research question and objectives: The primary objective of the study is to characterize and compare the risks of E4/DRSP with EE/DRSP and E4/DRSP with a pooled cohort of users of EE/LNG, EE/NETA, and EE/NGM combinations (non-DRSP-containing COCs) in a study population of actual users of these preparations under routine clinical practice. The main clinical outcome of interest is VTE. Secondary objectives include measuring the occurrence of unintended pregnancy, assessing the risk of ATE, deep venous thrombosis (DVT) of the lower extremities, and pulmonary embolism (PE), describing the drug utilization pattern, and describing the baseline risk for VTE and ATE.

Study design: The INAS-SEECS study is a comparative, prospective, active surveillance study that follows three cohorts. The cohorts consist of new users (starters and restarters ) of hormonal contraceptives and focus on two co-primary comparisons: E4/DRSP versus EE/DRSP and E4/DRSP versus non-DRSP COCs. The study uses a non-interventional approach to provide comprehensive information on these treatments in a routine clinical practice setting. Study participants will be enrolled via an international network of COC-prescribing health care professionals (HCPs) and followed up for two years. All outcomes of interest will be captured by direct contact with the study participants. Reported outcomes of interest will be validated via attending physicians and/or relevant source documents. The classification of outcomes of interest into 'confirmed' and 'not confirmed' will be verified by blinded independent adjudication.

Population: Approximately 68,100 study participants (22,700 E4/DRSP, 22,700 EE/DRSP, and 22,700 EE/LNG, EE/NETA, and EE/NGM users) will be recruited via a network of COC-prescribing HCPs in the USA. All new users (starters and restarters with at least two months break) prescribed E4/DRSP, EE/DRSP, EE/LNG, EE/NETA, or EE/NGM who are willing to participate may be eligible for enrollment in the study. The distribution of body mass index (BMI) categories will be monitored during the recruitment period, and if necessary, a quota will be introduced. However, women who have given birth six weeks before treatment starts will be excluded from the study. Participants with a prior cancer diagnosis (less than six months) and a prior VTE (Medical history of VTE at study entry) and those using anticoagulants will be excluded from the primary analysis of VTE. However, they will be considered in the sensitivity analyses.

Variables: The variable to determine the primary endpoint is the occurrence of a new VTE during follow-up. Two co-primary comparisons will be investigated; between E4/DRSP versus EE/DRSP and between E4/DRSP versus non-DRSP COC users. Variables to determine the secondary endpoints include the occurrence of ATE, DVT of the lower extremities, PE, and unintended pregnancies. Variables to characterize the baseline risk profile of users are baseline population characteristics, including BMI and smoking status, socio-economic factors, concomitant medication, and reproductive, contraceptive, and medical histories.

Data sources: The INAS-SEECS is a field study that entails exposure to COCs and the occurrence of clinical outcomes of interest by completing questionnaires at baseline (study entry) and follow-up (at 6, 12, 18, and 24 months post-baseline), in addition to potential confounding factors and potential effect modifiers. Study participants will be sent a reminder email at three and nine months to enhance the accuracy of self-reported information. Medical confirmation of the occurrence of a clinical outcome of interest will be sought from the attending HCP and/or study participant (e.g., diagnostic report, discharge letter).

Study size: The sample size calculation is based on an assumed incidence rate of nine VTE per 10,000 women-years (WY) for EE/DRSP and nine VTE per 10,000 WY for EE/LNG, EE/NETA, and EE/NGM. A total of 68,100 women (22,700 E4/DRSP users, 22,700 EE/DRSP users, and 15,000 EE/LNG users plus 7,700 EE/NETA and EE/NGM users) will be recruited within three years and followed up for two years considering treatment adherence, treatment stopping/switching, and lost-to-follow-up (LTFU)/dropout at a rate of 20%. Sample size calculations show that approximately 109,000 WY of observation is statistically sufficient (power=80%, α=0.025 one-sided, allocation rate 1:1) to exclude a 2.0-fold VTE risk for E4/DRSP users compared to users of EE/DRSP and for E4/DRSP users compared to users of non-DRSP COCs (i.e., EE/LNG, EE/NETA and EE/NGM).

Data analysis: The final analyses will include both an "as-treated" (AT) and an "intention-to-treat" (ITT) analysis. All eligible women will be assigned to the ITT and AT population at baseline. Only women with follow-up information will be considered for longitudinal analysis. Women who never started their prescribed baseline medication will be considered in the ITT analysis but excluded from the AT analysis. Population characteristics, e.g., socio-economic factors, parameters of reproductive, contraceptive history, and medical history, will be summarized descriptively and used to estimate the probability of treatment differences. A Marginal Structural Cox Model (MSM) with Inverse Probability Weighting (IPW) of treatment and censoring will be applied for the primary analysis. Hazard ratios for the VTE risk will be provided with corresponding 95% confidence intervals. Non-Inferiority of E4/DRSP will be concluded if the upper confidence limit for the point estimate of the adjusted VTE hazard ratio (HRVTE) is below the predefined non-inferiority limit of HRni=2 for both comparisons (HR for E4/DRSP vs. EE/DRSP AND E4/DRSP vs. non-DRSP COCs is less 2.0). If non-inferiority of E4/DRSP could be demonstrated, superiority to EE/DRSP or non-DRSP COCs will be subsequently evaluated.

Milestones: The INAS-SEECS study is expected to start in 12/2023 after the FDA approval of the protocol. The final study report will be available in 12/2029.

ELIGIBILITY:
Inclusion Criteria:

• New users of E4/DRSP or EE/DRSP or EE/LNG or EE/NGM or EE/NETA

Exclusion Criteria:

• Women who have given birth six weeks before treatment starts will be excluded from the study.

Sex: Female
Age Groups: Child, Adult, Older Adult
Study Population: Approximately 68,100 study participants (22,700 E4/DRSP, 22,700 EE/DRSP, and 22,700 EE/LNG, EE/NETA, and EE/NGM users) will be recruited via a network of COC-prescribing HCPs in the USA.
Sampling Method: Non-Probability Sample
Enrollment: 68100 (Estimated)
Dates: Start 2025-04-24 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2029-06 (Estimated)

PRIMARY OUTCOMES:
Co-primary endpoint considering the time-to-VTE event, specifically: New VTE | Up to 24 months post baseline
  ICD-10 codes: I80.1, I80.2, I80.3, I80.8*, I80.9, I81, I82.0, I82.2, I82.3, I82.8, I82.9, I26.*, I63.6, I67.6, H34.8, K55.0, N28.0
  The variable to determine the primary endpoint is:
  The average treatment effect is quantified as the hazard ratio (HR) of E4/DRSP to EE/DRSP and E4/DRSP to non-DRSP COCs. VTE events are measured as the occurrence (or absence) of a new (non-recurrent) confirmed VTE during follow-up.

SECONDARY OUTCOMES:
Incidence rate and time-to-event of ATE, including acute myocardial infarction | Up to 24 months post baseline
  AMI; ICD-10 code I21.*) and cerebrovascular accidents (CVA; ICD-10 code: I24.9, G45.*, I61.*, I63.1, I63.2, I63.3, I63.4, I63.5, I63.8, I63.9
Incidence rate and time-to-event of deep venous thrombosis (DVT) of the lower extremities | Up to 24 months post baseline
  ICD-10 codes: I80.1 and I80.2
Incidence rate and time-to-event of pulmonary embolism (PE) | Up to 24 months post baseline
  ICD-10 code: I26.*
Incidence rate and time-to-event of VTE and ATE, stratified analyses | Up to 24 months post baseline
  Stratification by age, smoking, BMI, and COC user status [first-time users and restarter])
Incidence rate and time-to-event of discontinuation/switching | Up to 24 months post baseline
Incidence rate and time-to-event of unintended pregnancy | Up to 24 months post baseline

CONTACTS AND LOCATIONS:
Overall Officials: Klaas Heinemann, Dr., Principal Investigator — ZEG Berlin GmbH
Locations (1):
- Berlin Center for Epidemiology and Health Research, Berlin, State of Berlin, Germany